CLINICAL TRIAL: NCT00277472
Title: A 28-week, Multicenter Study to Evaluate the Effects of Valsartan/Hydrochlorothiazide (160/12.5 mg) in Comparison With Hydrochlorothiazide (25 mg) Monotherapy, for the Treatment of Patients With Hypertension, Uncontrolled by Hydrochlorothiazide (12.5 mg) Monotherapy
Brief Title: Efficacy and Safety of Valsartan/Hydrochlorothiazide Combination Therapy in Patients With Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Study Director, Novartis Pharma
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAH631BUS04
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2008-03

CONDITIONS: Hypertension
Keywords: Hypertension; High blood pressure; diuretics; valsartan
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide; Water

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- valsartan HCTZ (Experimental)
  Interventions: Drug: Valsartan/Hydrochlorothiazide
- HCTZ (Active Comparator)
  Interventions: Drug: HCTZ

INTERVENTIONS:
Drug: Valsartan/Hydrochlorothiazide — 160/12.5 mg taken once daily orally
  Other Names: Co-Diovan, Diovan HCT
  Arms: valsartan HCTZ
Drug: HCTZ — 25 mg taken once daily orally
  Other Names: hydrochlorothiazice, water pill
  Arms: HCTZ

SUMMARY:
This study will assess the efficacy and safety of valsartan/hydrochlorothiazide combination therapy in patients with hypertension not controlled with hydrochlorothiazide monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age and older
* Diagnosed as having hypertension (mean seated systolic blood pressure ≥ 150 mm Hg but < 180 mm Hg and mean seated diastolic blood pressure ≥ 95 mm Hg and <110 mm Hg

Exclusion Criteria:

* - Patients with sever hypertension: Systolic ≥ 180 mm Hg or Diastolic ≥ 110 mm Hg
* Diabetes with fasting glucose > 126 mg/dl or on existing anti-diabetic medication
* History of stroke, transient ischemic attack, or myocardial infarction within the last 6 months, or diagnosed with congestive heart failure.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-11; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Blood pressure control (systolic blood pressure <140 and diastolic blood pressure <90mmHg) after 4 weeks
Blood pressure control (systolic blood pressure <140 and diastolic blood pressure <90mmHg) after 2 weeks and 20 weeks

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure after 2 weeks and 4 weeks
Change from baseline in diastolic blood pressure after 2 weeks and 4 weeks
Change in systolic blood pressure at 20 weeks compared to 4 weeks
Change in diastolic blood pressure at 20 weeks compared to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis 862-778-8300 Pharmaceuticals, Study Director — Novartis
Locations (1):
- Novartis, East Hanover, New Jersey, United States

REFERENCES:
- See also: Click here for more information about this study. — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?t=i&trialID=491&diseaseID=28